CLINICAL TRIAL: NCT00947479
Title: Effect of Correction of Obstructive Sleep Apnea With Positive Airway Pressure on Central Blood Pressure and Kidney and Endothelial Function
Brief Title: Effect of Obstructive Sleep Apnea on Central Blood Pressure and Kidney and Endothelial Function
Acronym: OSA-AKI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Lodz (Other)
Responsible Party: Professor Michał Nowicki, Department of Nephrology, Hypertension and Kidney Transplantation
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: UMLodz OSA-AKI
Record Dates: First submitted 2009-07-27; First posted 2009-07-28 (Estimated); Last update posted 2009-07-28 (Estimated); Status verified 2009-07

CONDITIONS: Obstructive Sleep Apnea; Acute Kidney Failure; Chronic Kidney Disease
Keywords: obstructive sleep apnea; pulse-wave velocity,; acute kidney injury; biomarkers of acute kidney injury
MeSH Terms: conditions — Sleep Apnea, Obstructive; Acute Kidney Injury; Renal Insufficiency, Chronic | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- continuous positive airway pressure (CPAP) (Other): CPAP will be applied in all patients
  Interventions: Other: continuous positive airway pressure (CPAP)

INTERVENTIONS:
Other: continuous positive airway pressure (CPAP) — After being qualified into the study according to the aforementioned inclusion criteria and after giving an informed consent the polysomnography will be performed in all patients during night rest.In all patients eligible to sleep apnea treatment according to apnea/hypopnea index (AHI, number of apneic/hypopneic episodes per 1 h of effective sleep) from diagnostic polysomnography, CPAP treatment will be introduced under polysomnographic surveillance and the same panel of clinical and biochemical parameters will be evaluated.
  Other Names: Epworth sleepiness scale (ESS)

SUMMARY:
Obstructive sleep apnea (OSA) is a frequently underdiagnosed condition that has emerged as an increasing medical problem with important social and financial implications worldwide. OSA is a well established risk factor for systemic hypertension myocardial infarction or stroke and it has been documented that blood pressure rises in a very consistent fashion during apneic episodes. The incidence of the episodes of apnea during sleep causes repeated subclinical acute kidney injuries (AKI) contributing to the development of CKD. One of the mechanisms responsible for AKI might be endothelial injury followed by an increase of central aortic pressure.

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) is a frequently underdiagnosed condition that has emerged as an increasing medical problem with important social and financial implications worldwide. Its prevalence may reach 25% in middle-aged men and 11% in women. The most important risk factor for OSA is obesity - every 10% weight gain increases the incidence of the disease 6 times. OSA usually occurs in middle age males and is characterized by history of snoring, daytime somnolence and nocturnal choking or gasping. The underlying cause is transient cessation of airflow due to occlusion of the oropharyngeal tract. Episodes of apnea are considered important if they persist for longer than 10 seconds, but in some cases they may last as long as 2 minutes. The airway occlusion results in recurrent hypoxia, hypercapnia, arousals from sleep, compensatory hyperventilation leading to secondary hypocapnia and generation of exaggerated negative intrathoracic pressure that all can either directly or indirectly be harmful to the cardiovascular system through several pathways like sympathetic activation, inflammation, oxidative stress and endothelial dysfunction. Recurrent episodes of apnea/hypoxia may negatively affect the function of many organs, e.g. they induce (cyclical bradycardia during the apneic episodes, followed by tachycardia during the ensuing ventilatory phases) or rise blood pressure. Moreover, OSA is a well established risk factor for systemic hypertension myocardial infarction or stroke and it has been documented that blood pressure rises in a very consistent fashion during apneic episodes. The mechanisms responsible for this phenomenon are complex because the direct effects of apnea (hypoxemia and low intrathoracic pressure) are modified by cardiopulmonary reflexes. Undoubtedly, the rapid increase in arterial pressure that occurs at the end of an apneic episode is mainly mediated by surges in sympathetic function during the arousal reaction.

Hypertension has emerged as a second, after diabetes mellitus, most frequent cause of chronic kidney disease (CKD). The rise of arterial blood pressure and endothelial damage due to ischaemia during apneic episodes may contribute to CKD. According to the recent findings OSA patients are much more frequently diagnosed with chronic kidney disease. The high frequency of OSA in patients with renal function impairment could be explained by the fact that the most common comorbid conditions of CKD, namely atherosclerosis and diabetes, are also independently associated with his syndrome. The detailed pathogenesis of the strong relation between OSA and CKD has not been investigated so far.

OSA patients are characterized by arterial stiffness, evaluated by pulse-wave velocity (PWV). PWV is a sensitive and validated marker of cardiovascular risk, including premature coronary artery disease, atherosclerosis, stroke and cardiovascular mortality.

The diagnosis of acute kidney injury (AKI) is routinely based on changes in serum creatinine, but its measurements are a poor indicator of acute deterioration in kidney function. First, serum creatinine concentrations might not change until about 50% of kidney function has already been lost. Second, serum creatinine levels can vary widely with age, sex, muscle mass, muscle metabolism, medications and hydration status. Novel, more specific and sensitive biomarkers of AKI are neutrophil gelatinase-associated lipocalin (NGAL), cystatin C, kidney injury molecule 1 (KIM-1), liver-type fatty acid-binding protein (L-FABP), which concentrations in both urine or serum rise significantly in patients with AKI and correlate with severity of kidney injury.

CKD is a devastating illness that has reached epidemic proportions worldwide. CKD is characterized by a progressive decline in kidney function that is associated with excess morbidity and mortality. The deterioration of kidney function can be delayed and patient outcome favorably affected if kidney disease is recognized and treated in a timely manner.

In our study we would like to prove that apneic episodes during sleep can cause repeated renal ischaemia-reperfusion injuries, which may lead to repeated acute subclinical kidney injuries (AKI) contributing to the development of chronic kidney disease.

The aim of this project is to study the influence of sleep apnea syndrome on the markers of acute kidney injury, endothelial function, arterial stiffness and central aortic pressure.

ELIGIBILITY:
Inclusion Criteria:

1. Males with high risk of obstructive sleep apnea syndrome as clinically assessed by coincidence of typical symptoms (e.g. daily somnolence, witnessed apnea, non-refreshing sleep), obesity and high score on Epworth sleepiness scale (ESS) with age range from 18 to 70 years
2. Glomerular filtration rate (MDRD formula-based) > 60 ml/min
3. Arterial hypertension diagnosed according to the European Society of Hypertension 2007 Guidelines.

Exclusion Criteria:

1. Mental illness
2. Proteinuria >2 g/24h
3. Acute and chronic inflammation
4. Heart failure III or IV grade
5. Uncontrolled diabetes mellitus
6. Severe lipid disturbances (triglyceride and/or total cholesterol concentration > 300 mg/dl)
7. Chronic administration of drugs with confirmed nephrotoxicity and/or sympathicomimetics
8. Obstructive and restrictive pulmonary diseases which may deteriorate the function of the respiratory system

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2009-02; Primary Completion 2010-06 (Estimated); Study Completion 2011-07 (Estimated)

PRIMARY OUTCOMES:
presence of acute kidney injury | one year

CONTACTS AND LOCATIONS:
Overall Officials: Michał Nowicki, MD, PhD, Study Chair — Medical University of Lodz, Poland
Locations (1):
- Medical University, Lodz, Łódź Voivodeship, Poland